CLINICAL TRIAL: NCT04694274
Title: Genetic Polymorphisms and Their Association With Temporomandibular Disorders
Acronym: GenPolTMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Iva Alajbeg, Prof, University of Zagreb
Other Study IDs: IP-2019-04-6211
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Temporomandibular Disorders; Orofacial Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: patients with temporomandibular disorders
  Interventions: Device: stabilization splint; Procedure: physical therapy; Device: placebo splint
- group 2: healthy control

INTERVENTIONS:
Device: stabilization splint — The device made of a hard acrylic on stone cast of the upper jaw in the centric relation position. It has a thickness of 1.5 mm at the level of the first molar.
  Groups: group 1
Procedure: physical therapy — Home-exercise program included exercises for passive and active stretching, joint mobilization, passive extension, and translational movements to the right, left, and forward.
  Groups: group 1
Device: placebo splint — The placebo splint was made of thin heat-treatable foil (0.5 mm). The foil was heated and printed over a plaster model of the upper jaw resulting in a very thin film over the occlusal surfaces of all teeth.
  Groups: group 1

SUMMARY:
Temporomandibular disorders (TMD) are the most common orofacial pain disorders of non-dental origin with the prevalence of 6.1-10.2%, and incidence of 3.9%. Observable pathology is mostly absent, and the etiology often remains unknown. Since some other painful conditions of unknown origin (eg. fibromyalgia), also imply genetic factors, the aim of the study is to investigate genetic predisposition in relation to the risk for TMD onset. This will be achieved through analysis of polymorphisms in the selected genes in TMD patients (DC/TMD) and matched control subjects. The possibility of involvement of specific polymorphisms in modulation of therapy response will also be investigated. The hypotheses: (I) the Single Nucleotide Polymorphism (SNPs) clustering will be dependent on presence or absence of TMD (comparison of patients with control subjects), and will possibly depend on source of pain, pain intensity, presence of bone changes, psychological features and previous orthodontic therapy, and (II) SNPs will influence the treatment response. Along with anamnestic and clinical examination and occlusal splint therapy, genomic DNA will be analyzed from the buccal swabs. Isolated DNA will be used for the determination of 19 polymorphisms of selected genes using Real-Time PCR method. The analysis of salivary oxidative stress markers and opiorphin will be also performed, as their relationship with TMD has been shown previously. This time, their concentration will be associated with polymorphisms in the promoters of genes responsible for their synthesis. The investigators expect to show that particular gene profile or group of SNPs represent a risk factor for TMD development. Innovative approach of the concept of determining the genetic predisposition for TMD has the potential for development of commercial genetic test with potential for risk estimation in relation to TMD onset. This could enable early interventions and active avoidance of environmental risk factors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of myofascial pain / arthralgia / painful disc displacement according to Diagnostic Criteria for Temporomandibular Disorders (DC/TMD)
* average pain in the last 10 days >30 mm on a Visual Analogue Scale
* pain duration of at least 3 months
* good oral hygiene
* presence of own natural teeth
* absence of any form of chronic pain in the orofacial region or in other regions of the body

Exclusion Criteria:

* other orofacial pain conditions including dental pain
* poor oral hygiene, gingivitis or periodontitis
* chronic medical conditions (diabetes, cardiovascular diseases, cancer, and autoimmune diseases) - - -
* neurological and psychiatric disorders
* pregnancy
* causes of headache, unrelated to TMD, listed in the International Classification of Headache Disorders

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will include subjects, 15 years and older, with a report of ongoing for a duration of >3 months and diagnosis of TMD according DC/TMD and age matched control subjects
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline characteristic pain intensity at 6 months | baseline, 6th month
  The characteristic pain intensity (part of Graded Chronic Pain Scale, GCPS) compute mean of items (pain right now, worst pain, average pain), and multiply by 10.
  Each item ranges from 0 to 10, with higher scores mean a worse outcome.
change from baseline spontaneous pain at 6 months | baseline, 6th month
  For evaluation of spontaneous pain from the temporomandibular joint and the masticatory muscles a 100 mm horizontal Visual analogue scale (VAS) is used. Visual analogue scale ranges from 0 to 100, with higher scores mean a worse outcome.

SECONDARY OUTCOMES:
change from baseline range of mouth opening at 6 months | baseline, 6th month
  1. The pain-free opening is defined as the maximum amount that a patient achieves by opening the mouth without feeling pain and is measured as the distance between the incisal edges of the upper and lower central incisors.
  2. Maximum unassisted mouth opening is measured as the distance between the maxillary and mandibular central incisors and defined as the largest amount of opening that a patient can achieve regardless of pain and discomfort.
change from baseline anxiety at 6 months | baseline, 6th month
  the General anxiety disorder questionnaire (GAD-7) (a 7-question questionnaire that assesses the severity of respondents' anxiety symptoms) is used for assessing the severity of anxiety symptoms of the participants. Scale ranges fro 0 to 21, with higher scores mean a worse outcome. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.
change from baseline depression at 6 months | baseline, 6th month
  The Patient Health Questionnaire-9 (PHQ-9) is used for measuring the severity of depressive symptoms. Scores range from 0 to 27, with cut-points 5, 10, 15, and 20 represent mild, moderate, moderately severe and severe depression, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Iva Z Alajbeg, Principal Investigator — School of Dental Medicine, University of Zagreb
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, N/A = Not Applicable, Croatia

REFERENCES:
- [Background] Alajbeg IZ, Lapic I, Rogic D, Vuletic L, Andabak Rogulj A, Illes D, Knezovic Zlataric D, Badel T, Vrbanovic E, Alajbeg I. Within-Subject Reliability and between-Subject Variability of Oxidative Stress Markers in Saliva of Healthy Subjects: A Longitudinal Pilot Study. Dis Markers. 2017;2017:2697464. doi: 10.1155/2017/2697464. Epub 2017 Nov 15. PMID 29269980
- [Background] Vrbanovic E, Alajbeg IZ. Long-term Effectiveness of Occlusal Splint Therapy Compared to Placebo in Patients with Chronic Temporomandibular Disorders. Acta Stomatol Croat. 2019 Sep;53(3):195-206. doi: 10.15644/asc53/3/1. PMID 31749451
- [Background] Vrbanovic E, Lapic I, Rogic D, Alajbeg IZ. Changes in salivary oxidative status, salivary cortisol, and clinical symptoms in female patients with temporomandibular disorders during occlusal splint therapy: a 3-month follow up. BMC Oral Health. 2019 Jun 6;19(1):100. doi: 10.1186/s12903-019-0791-8. PMID 31170954
- [Background] Vrbanovic E, Alajbeg IZ, Vuletic L, Lapic I, Rogic D, Andabak Rogulj A, Illes D, Knezovic Zlataric D, Badel T, Alajbeg I. Salivary Oxidant/Antioxidant Status in Chronic Temporomandibular Disorders Is Dependent on Source and Intensity of Pain - A Pilot Study. Front Physiol. 2018 Oct 17;9:1405. doi: 10.3389/fphys.2018.01405. eCollection 2018. PMID 30386251
- [Background] Alajbeg IZ, Gikic M, Valentic-Peruzovic M. Mandibular Range of Movement and Pain Intensity in Patients with Anterior Disc Displacement without Reduction. Acta Stomatol Croat. 2015 Jun;49(2):119-27. doi: 10.15644/asc49/2/5. PMID 27688394
- [Result] Alajbeg IZ, Vrbanovic E, Lapic I, Alajbeg I, Vuletic L. Effect of occlusal splint on oxidative stress markers and psychological aspects of chronic temporomandibular pain: a randomized controlled trial. Sci Rep. 2020 Jul 3;10(1):10981. doi: 10.1038/s41598-020-67383-x. PMID 32620810
- [Result] Vrbanovic E, Alajbeg IZ, Alajbeg I. COVID-19 pandemic and Zagreb earthquakes as stressors in patients with temporomandibular disorders. Oral Dis. 2021 Apr;27 Suppl 3(Suppl 3):688-693. doi: 10.1111/odi.13488. Epub 2020 Jul 13. PMID 32533874
- [Derived] Alajbeg IZ, Vrbanovic E, Alajbeg I, Orabovic I, Naka K, Mrla A, Boucher Y. Time-course of pain and salivary opiorphin release in response to oral capsaicin differ in burning mouth syndrome patients, temporomandibular disorders patients and control subjects. Clin Oral Investig. 2024 Apr 9;28(5):246. doi: 10.1007/s00784-024-05653-y. PMID 38589630
- [Derived] Vrbanovic E, Zlendic M, Alajbeg IZ. Association of oral behaviours' frequency with psychological profile, somatosensory amplification, presence of pain and self-reported pain intensity. Acta Odontol Scand. 2022 Oct;80(7):522-528. doi: 10.1080/00016357.2022.2042380. Epub 2022 Mar 7. PMID 35254961
- [Derived] Gikic M, Vrbanovic E, Zlendic M, Alajbeg IZ. Treatment responses in chronic temporomandibular patients depending on the treatment modalities and frequency of parafunctional behaviour. J Oral Rehabil. 2021 Jul;48(7):785-797. doi: 10.1111/joor.13173. Epub 2021 Apr 12. PMID 33797785